CLINICAL TRIAL: NCT05303493
Title: Phase I Trial of Camu Camu Prebiotic and Immune Checkpoint Inhibition in Patients With Non-Small Cell Lung Cancer and Melanoma
Brief Title: Camu-Camu Prebiotic and Immune Checkpoint Inhibition in Patients With Non-small Cell Lung Cancer and Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21.393
Record Dates: First submitted 2021-09-22; First posted 2022-03-31 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage IV; Melanoma Stage IV; Unresectable Melanoma; Advanced Non-Small Cell Lung Cancer
Keywords: CamuCamu; Prebiotics; Immune check points
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Intervention Model Description: Cohort 1. For patients with advanced NSCLC, treatment will consist of ICI in combination with CamuCamu.
  Cohort 2. For patients with advanced cutaneous melanoma, treatment will consist of single-agent anti-PD-1 either nivolumab or pembrolizumab at the discretion of the treating physician in combination with investigational CC capsules Cohort 3. For patients with advanced melanoma receiving standard-of-care ICI who exhibit either an ORR of SD or PD during the first 3 months of ICI initiation, their current regimen will continue unchanged and they will receive Camu C and will be continued for 18 weeks or upon progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camu-camu (intervention) in addition to standard-of-care ICI (Experimental): Camu-camu (intervention) will be added to standard-of-care ICI in:
  Cohort 1. For patients with advanced NSCLC, treatment will consist of single-agent pembrolizumab in combination with physician's choice platinum-doublet chemotherapy in combination with CC.
  Cohort 2. For patients with advanced cutaneous melanoma, treatment will consist of single-agent anti-PD-1 either nivolumab or pembrolizumab at the discretion of the treating physician.
  Cohort 3. For patients with advanced melanoma receiving standard-of-care ICI (either single-agent anti-PD-1 or combination anti-CTLA-4 plus anti-PD-1) who experience progressive disease (PD), their current regimen will continue unchanged and they will receive CC at 1500 mg for 3 months or until confirmed progression if progression occurs earlier.
  Interventions: Biological: Camu Camu Capsules (Camu Camu powder encapsulated (500mg each) + ICI

INTERVENTIONS:
Biological: Camu Camu Capsules (Camu Camu powder encapsulated (500mg each) + ICI — Evaluate the safety and tolerability of CC prebiotic in addition to ICI in patients with NSCLC and melanoma

SUMMARY:
Modulating the gut microbiome to improve response to immune-checkpoint inhibitors is an active area of study. Prebiotic substances (compounds which positively shift the gut microbiome) are a reliable and safe method of gut microbiome modulation. Data suggest that the berry Camu Camu (CC), also known as Myrciaria dubia has prebiotic potential to enrich Akkermansia muciniphila, a bacterium shown to alleviate metabolic disorders and improve ICI efficacy in preclinical models. Our primary objective is to assess the safety and tolerability of CC prebiotic in patients with advanced NSCLC and melanoma in combination with standard-of-care ICI.

DETAILED DESCRIPTION:
Immune-checkpoint inhibitors (ICI) now represent the backbone therapy for patients with advanced or unresectable non-small cell lung cancer (NSCLC) and metastatic melanoma. However, only a minority of patients obtain durable complete responses.

In patients with advanced NSCLC with a Programmed Death Ligand-1 (PD-L1) expression level below 50%, the standard-of-care is pembrolizumab plus platinum doublet chemotherapy, with overall survival (OS) at 2 years reaching 46%. In patients with advanced melanoma, combination of anti-CTLA-4 (ipilimumab) and anti-PD-1 (nivolumab) is a key standard-of-care option. In a study in patients with advanced melanoma evaluating the combination regimen of nivolumab plus ipilimumab group, OS at 5 years was 52% in the nivolumab plus ipilimumab group and 44% in the nivolumab group, as compared with 26% in the ipilimumab group.

Despite these improvements in outcomes with ICI, these survival and response rates remain suboptimal, and therefore, developing strategies to safely increase ICI efficacy or reverse ICI resistance represents an unmet clinical need. Moreover, there are currently no available options for patients who progress on standard-of-care ICI. Recent pre-clinical studies have demonstrated the role of the gut microbiome in improving ICI efficacy, and therefore, efforts to modulate the gut microbiome is an active area of study. Indeed, two phase I clinical studies evaluating gut microbiome modulation with fecal microbial transplantation (FMT) demonstrated increase in objective response rate compared to historical controls. Moreover, studies in over 8,000 patients (including patients with NSCLC and melanoma) have confirmed the independent and negative role of antibiotics (ATB) in patients receiving ICI, further validating the important role of the gut microbiome.

Therefore, it is clear that modulation of the gut microbiome represents a promising therapeutic strategy in improving ICI efficacy. Other than FMT, prebiotic substances (compounds which positively shift the gut microbiome) are a reliable and safe method of gut microbiome modulation. Data suggest that the berry Camu Camu (CC), also known as Myrciaria dubia has prebiotic potential to enrich Akkermansia muciniphila, a bacterium shown to alleviate metabolic disorders and improve ICI efficacy in preclinical models. Our preclinical work showed that CC oral supplementation significantly decreased tumor size and had an additive effect in combination with anti-PD-1 in two murine tumor models, MCA-205 (anti-PD-1 sensitive) and E0771 (anti-PD-1 resistant). Flow cytometry and RNA seq analysis of the tumor microenvironment (TME) and T cell depletion showed that CC's anti-tumor effect was dependent on CD8+ T cells. Moreover, CC supplementation was able to transform an anti-PD-1-resistant tumor into an anti-PD-1-sensitive tumor. ATB administration inhibited CC activity, proving that the activity of CC was dependent on the gut microbiome. The 16S rRNA profiling of murine fecal samples showed that CC increased bacterial diversity and enrichment of beneficial bacteria.

CC is available over the counter as a natural prebiotic and has been approved for human clinical trials in obesity (NCT04130321) and HIV (NCT04058392).

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent;
2. Age 18 years or older;
3. One of the following histological-confirmed diagnoses**
4. No prior anti-PD1 treatment (except for patients in cohort 3)
5. Evaluable disease as per RECIST 1.1;
6. ECOG performance status of 0-2;
7. Ability to ingest capsules;
8. Patients receiving systemic steroids at physiologic doses are permitted to enroll provided the dose not exceed 10 mg prednisone daily or equivalent;
9. Negative pregnancy test for women of child-bearing potential; and
10. Highly effective contraception (any method above 97% success rate) for both male and female subjects throughout the study and for at least 60 days after last treatment administration, if the risk of conception exists

    * a.Cohort 1: patients with stage IV or unresectable NSCLC (including squamous cell carcinoma) with PD-L1 expression <50% who are going to be treated with anti-PD-1 in combination with platinum-doublet chemotherapy b.Cohort 2: Patients with untreated stage IV or unresectable cutaneous melanoma, acral or mucosal melanoma who are going to be treated with single-agent anti-PD-1 therapy i. Patients with prior treatment with BRAF-targeting agents (BRAF inhibition +/- MEK inhibition) are permitted to enroll ii. Patients with melanoma of unknown primary are permitted to enroll. Diagnosis of melanoma of unknown primary at the discretion of the treating oncologist and sponsor c.Cohort 3: Patients with stage IV or unresectable cutaneous melanoma, acral or mucosal melanoma already receiving standard-of-care ICI (either single-agent anti-PD-1 or combination anti-CTLA-4 plus anti-PD-1) at the first sign of progression i.Patients with melanoma of unknown primary are permitted to enroll. Diagnosis of melanoma with unknown primary at the discretion of the treating oncologist and PI.

Exclusion criteria

1. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment;
2. Has a diagnosis of severe immunodeficiency (e.g. transplantation) or receiving systemic steroid therapy (>10mg prednisone daily or equivalent) or any other form of active immunosuppressive therapy at the discretion of the sponsor;

   a. Patients with well-controlled HIV who are on HAART and have undetectable viral load are permitted to enroll;
3. Use of probiotics. Probiotics must be discontinued a minimum of 2 weeks before CC administration and patients are not permitted to take probiotics during the course of immunotherapy treatment;
4. Use of natural supplements including prebiotics. Prebiotics must be discontinued a minimum of 2 weeks before CC administration and patients are not permitted to take other prebiotics during the course of immunotherapy treatment;
5. Use of antibiotics within 2 weeks of enrollment in the study;

   a. If a patient requires antibiotics during CC treatment, they are permitted to stay on the study.
6. Expected to require any other form of systemic anti-neoplastic therapy while on study (radiation therapy is permitted);
7. In the last year, has a known history of a malignancy requiring anti-neoplastic treatment.

   a. NOTE: This time requirement does not apply to patients who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cancers including cervical cancer, breast cancer, melanoma, or other in situ cancers;
8. Symptomatic central nervous system (CNS) metastases
9. Leptomeningeal involvement (leptomeningeal enhancement on MRI/CT imaging and/or positive CSF cytology);
10. Has an uncontrolled autoimmune disease that requires systemic steroids or immunosuppressive agents;

    a. Patients with vitiligo, type I diabetes, well controlled hypothyroidism due to Hashimoto disease, resolved childhood asthma/atopy are permitted to enroll.
11. A history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
12. Has serious concomitant illnesses, such as: impaired cardiovascular function or clinically significant cardiovascular disease (uncontrolled congestive heart failure requiring treatment (NYHA grade > 3), uncontrolled hypertension, acute myocardial cardiac ischemia or unstable angina < 2 months prior to study entry, and severe cardiac arrhythmia), active inflammatory bowel disorders.
13. Active kidney disease/severe chronic kidney or liver disease or hematological blood test alteration that would preclude safe administration of chemotherapy at the discretion of the sponsor.
14. Has an active infection requiring systemic therapy;
15. Patient has received a live vaccine within 4 weeks prior to the first dose of treatment

    a. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed. COVID-19 vaccinations are not live vaccinations and are allowed.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
17. Known life-threatening or severe allergy to CC at the discretion of the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (safety and tolerability) in patients with NSCLC and melanoma | At the end of every cycle (each cycle is 21 or 28 days, depending of the ICI treatment) until disease progression, then, every 3 months thereafter (for up to a total of 2 years)
  Safety of administration of CamuCamu in the Safety Analysis Dataset. The assessment of safety will be based on the incidence of AEs, SAEs, AEs leading to discontinuation, and deaths in the Safety Analysis dataset.
  Treatment-related adverse events will be graded according to the NCI CTCAE v5.0. of CC prebiotic in addition to ICI in patients with NSCLC and melanoma on the basis of the following endpoints:
  * Incidence and severity of AEs, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0)
  * Change from baseline in targeted vital signs
  * Change from baseline in targeted clinical laboratory test results

SECONDARY OUTCOMES:
Objective response rate in the NSCLC and melanoma cohort by RECIST criteria. | At 3 and 6 months, then at 12 months and up to 2 years
  To evaluate the preliminary activity of CC in combination with single-agent anti-PD-1 in patients with melanoma, and in combination with anti-PD-1 and chemotherapy in patients with advanced NSCLC as measured by ORR (ORR; the rate of complete response plus partial response, as per the iRECIST and RECIST criteria).
  Objective Response Rate (ORR) as defined by the proportion of patients with NSCLC and melanoma whose Best Overall Response (BOR) is either a complete response (CR) or partial response (PR) as assessed by iRECIST, based on RECIST v1.1. BOR is defined as the best response designation over the study as a whole, recorded between the dates of first dose until the last tumor assessment prior to subsequent therapy. CR or PR determinations included in the BOR assessment must be confirmed by a second scan performed no less than 4 weeks after the criteria for response are first met.

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Elkrief, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (3):
- Canada (3):
  - CISSS de la Montérégie-Centre- Hôpital Charles-Le Moyne, Longueuil, Quebec
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Pang SA, Elkrief A, Capella MP, Miller WH Jr. Two Cases of Durable and Deep Responses to Immune Checkpoint Inhibition-Refractory Metastatic Melanoma after Addition of Camu Camu Prebiotic. Curr Oncol. 2023 Aug 25;30(9):7852-7859. doi: 10.3390/curroncol30090570. PMID 37754485